CLINICAL TRIAL: NCT05776576
Title: Physical Activity and Recreation School Program for Special Needs Individuals With Physical Disabilities and Their Parents
Brief Title: Physical Activity and Recreation School Program for Special Needs Individuals and Their Parents
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Nilay Arman, Assoc. Prof., Istanbul University - Cerrahpasa
Other Study IDs: NAAArman
Record Dates: First submitted 2023-02-25; First posted 2023-03-20 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Adolescent Behavior; Children, Only; Child Behavior Problem
Keywords: Physical Inactivity; Physical Disability; Adolescent Behavior; Children, Only; Child Behavior Problem
MeSH Terms: conditions — Adolescent Behavior; Sedentary Behavior | interventions — Educational Status

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Special needs children and adolescents with physical disabilities and their parents: Project consists of three main stages as evaluation, education and experimentation. For evaluation, firstly physical activity levels of individuals with special needs, barriers in physical activity, and motivators will be determined with an interactive roundtable meeting with children, adolescents and their parents. Afterwards, posture analyzes of individuals with special needs will be performed by physiotherapists. For education, interactive informative seminars titled "Physical Activity in Individuals with Special Needs" will be given and after that posture and ergonomics education will be given to the participants individually. For experimentation, group exercises, dance therapy and technology-supported exercise educations will be implemented by physiotherapists, taking into account the previous evaluations.
  Interventions: Behavioral: Evaluation; Behavioral: Education; Other: Experimentation

INTERVENTIONS:
Behavioral: Evaluation — Within the scope of the evaluation, first of all, physical activity levels of children and adolescents with physical disabilities, barriers that prevent them from participating in physical activity, and motivators that can increase their participation will be determined, accompanied by an interactive roundtable meeting. Afterwards, posture analyzes of children and adolescents with special needs with physical disabilities will be performed by physiotherapists.
Behavioral: Education — In the education part, interactive informative seminars titled "Physical Activity in Individuals with Special Needs" will be given and after the objective posture assessments, postural disorders of children and adolescents with special needs will be determined and accordingly, posture and ergonomics training will be given to the participants individually.
Other: Experimentation — In the experimentation part, group exercises, dance therapy programs and technology-supported exercise educations with various technological equipment will be implemented in the company of physiotherapists, taking into account the posture assessments.

SUMMARY:
The general purpose of this project; "Physical Activity and Recreation School" for the evaluation of physical activity behaviors of individuals with physical disabilities between the ages of 6-18, to increase the level of knowledge and awareness of these individuals and their parents, and to enable individuals with special needs to experience sports activities in the company of health and sports professionals who are experts in their fields. is to arrange. This project consists of three main topics as evaluation, training and experimentation.

During the evaluation phase, interactive roundtable activity, valid and reliable scales and physical assessments, and barriers and motivators for physical activity participation of individuals with special needs will be evaluated. A comprehensive interactive training seminar on physical activity will be held for individuals with special needs and parents during the training phase.

In the experimentation phase, children and adolescents with special needs will participate in training programs that include exercise and sportive activities suitable for the determined physical activity barriers and motivators, and will have the opportunity to experience exercises and sportive activities that they have not experienced before. The results of this project will provide gains in the analysis and application of physical inactivity, which is seen as an important public health problem in our country, for individuals with special needs, and will also guide many relevant institutions, health professionals and educators.

ELIGIBILITY:
Inclusion Criteria:

For Individuals with special needs;

* Between the ages of 6-18
* Being diagnosed with Cerebral Palsy, Neuromuscular Muscle Disease, Spina Bifida or having a chronic neurological or orthopedic problem that causes physical disability
* Being in a wheelchair/ able to walk with an assistive device or independently
* Have a cognitive level to understand and communicate questions
* Being residing in the province of Istanbul For parents of individuals with special needs;
* Being the mother or father of a special needs child or adolescent
* Volunteering for a special needs child to participate in the study
* Being able to participate in the activities to be held within the scope of the project on a full-time basis
* Have a cognitive level to understand and communicate questions
* Using a smart phone.

Exclusion Criteria:

For Individuals with special needs;

* Having a cognitive problem that will prevent the application of the evaluation parameters
* Failure to approve the assessment by the custodial parent
* Having had lower extremity surgery in the last 6 months
* Doing regular physical activity in the last 6 months
* Being a professional athlete For parents of individuals with special needs;
* Being illiterate.
* Not living with a special needs child.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with special needs between the ages of 6-18 with physical disabilities and their families
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2023-01-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Observational Posture Analysis | Baseline
  Observational posture assessment will be made from the front, back and both sides of children and adolescents with physical disabilities while sitting or standing.
Physical Activity Participation Motivation Scale | Baseline
  The lowest score that can be obtained from the scale is 16, and the highest score is 80. The high scores of the participants on the scale mean that their motivation to participate in physical activity is positive.
Motivation Scale for Participation in Sports for Persons with Disabilities | Baseline
  The scale consists of 22 items and three sub-dimensions (intrinsic motivation, extrinsic motivation and amotivation). The scale, which was developed to reveal the sources of the motivations of the participants that cause them to do sports, is in the form of a 5-point Likert type. The answer options for the items in the 5-point Likert scale are "1=Strongly Disagree", "2=Partially Disagree", "3=Moderately Agree", "4=Agree", "5=Strongly Agree". Since the scores in the scale are between 1 and 5, the higher the propositions in the items, the higher the motivation level of students to participate in sports; The closer it is to 1, the lower it is considered.
Life Satisfaction Scale in Children | Baseline
  This scale consists of 5 questions in a 5-point Likert type (I strongly disagree 1, I strongly disagree 2, I am undecided 3, I somewhat agree 4, I completely agree 5) and it has a single factor structure.
Satisfaction Level | Change from Baseline Satisfaction Level at 3 months
  During and after the education, the level of satisfaction obtained by the parents thanks to the educational seminar will be evaluated with a 3-5 question questionnaire prepared by the project team. In addition, the satisfaction level of the participants will be evaluated with a numerical rating scale after each education and experimentation through Google Forms. This scale consists of numbers ranging from "0" to "10" points. Individuals will be asked to rate their satisfaction level with the best satisfaction level as "10" points and the worst satisfaction level with "0" points.
Level of Knowledge | Change from Baseline Level of Knowledge at 3 months
  During and after the education, the level of knowledge gained by the parents through the educational seminar will be evaluated with a 3-5 question questionnaire prepared by the project team. In addition, the knowledge level of the participants will be evaluated with a numerical rating scale after each education and experimentation through Google Forms. This scale consists of numbers ranging from "0" to "10" points. Individuals will be asked to rate their level of knowledge with the best knowledge level as "10" points and the worst knowledge level with "0" points.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc. Prof., Principal Investigator — Istanbul University-Cerrahpaşa, Department of Physiotherapy and Rehabilitation; İpek Yeldan, Prof., Study Chair — Istanbul University-Cerrahpaşa, Department of Physiotherapy and Rehabilitation; Asena Yekdaneh, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Elçin Akyürek, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education; İrem Kurt, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education; Tuğçe Poyraz, Pt., MSc., Study Chair — Istanbul University-Cerrahpasa Institute of Postgraduate Education
Locations (2):
- Turkey (Türkiye) (2):
  - Avcılar Belediyesi Gülten Nakipoğlu Engelli Yaşam Merkezi, Istanbul
  - Istanbul University-Cerrahpaşa Faculty of Health Sciences, Istanbul

IPD SHARING:
Plan to Share IPD: No